CLINICAL TRIAL: NCT06016478
Title: The Effect of 4 Weeks of L-Citrulline Supplementation on Macro- and Microvascular Function in Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Texas Tech University (Other)
Responsible Party: Principal Investigator, Arturo Figueroa, Arturo Figueroa, Principal Investigator, Texas Tech University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: IRB2022-1056
Record Dates: First submitted 2023-08-19; First posted 2023-08-29 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2023-10

CONDITIONS: Type 2 Diabetes
Keywords: Endothelial function; Arterial stiffness; Hyperglycemia; Oral glucose tolerance test; Aortic blood pressure; Blood glucose; Lean mass
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hyperglycemia | interventions — Citrulline

STUDY DESIGN:
Intervention Model Description: Double-blind (subject, investigator), randomized, cross-over, placebo-controlled
Who Masked: Participant, Investigator
Masking Description: Double-blind (subject, investigator), randomized, cross-over, placebo-controlled
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- L-citrulline (Experimental): 6 grams/day
  Interventions: Dietary Supplement: L-citrulline
- Placebo (Placebo Comparator): Microcrystalline cellulose
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: L-citrulline — 4 weeks of L-citrulline (6 g/day) in 8 capsules. Supplementation will be ingested daily, half of the doses in the morning and half at night.
  Arms: L-citrulline
Dietary Supplement: Placebo — 4 weeks of microcrystalline cellulose in 8 capsules. Supplementation will be ingested daily, half of the doses in the morning and half at night.
  Arms: Placebo

SUMMARY:
The purpose of this study is to examine the effect of 4 weeks of Citrulline supplementation on macro- and microvascular function during acute hyperglycemia in middle-aged and older adults with type 2 diabetes.

DETAILED DESCRIPTION:
Using a double-blind, randomized, placebo-controlled, and cross-over design, middle-aged and older adults with type 2 diabetes will be randomized to receive either CIT supplementation (6g/day) or placebo (Microcrystalline Cellulose, 6g/day) for 4 weeks.

There will be a total of 5 laboratory visits. Visit 1 (screening visit) will take approximately 1 hour and 30 minutes, visit 2 will take approximately 2 hours and 30 minutes, and visits 3-5 will be approximately 3 hours each.

Visit 1 will measure blood pressure, blood glucose and lipid levels, anthropometry, body composition, and muscle strengths. Visits 2-5 will assess vascular function and glucose control during fasted and acute hyperglycemia conditions induced by 75g of glucose ingestion.

ELIGIBILITY:
Inclusion Criteria:

* Middle-aged and older women and men between 40-75 years old
* A physician diagnosed type 2 diabetes at least 3 months ago
* Treated with an oral hypoglycemic medication
* Body mass index < 40 kg/m2
* Systolic blood pressure < 160 mmHg
* Sedentary (defined as < 120 min/week of exercise)
* Not currently participating in exercise or dietary interventions for at least 2 months prior the present study and willing to abstain from participating in those strategies during the duration of this study.

Exclusion Criteria:

* < 40 years of age and > 65 years of age
* Use of medications and/or any supplements that may affect outcome variables (such as arginine- or citrulline-containing supplements, nitrates, and nitroglycerin)
* Body mass index ≥ 40 kg/m2
* Systolic blood pressure ≥ 160 mmHg
* Recent changes in medications within 3 months
* Current smoking any tobacco use
* Type 1 diabetes, severe cardiovascular/renal/pulmonary diseases
* More than 7 alcoholic drinks/week of consumption
* Premenopausal women with an irregular menstrual cycle (oligomenorrhea) or pregnancy

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
Change in macrovascular endothelial function in the fasted condition | 4 weeks
  Macrovascular endothelial function will be measured using brachial artery flow mediated dilation (ultrasonography) during reactive hyperemia at baseline and after 4 weeks of supplementation.
Change in macrovascular endothelial function during acute hyperglycemia | 4 weeks
  Macrovascular endothelial function will be measured using brachial artery flow mediated dilation (ultrasonography) during reactive hyperemia at 60 minutes after oral glucose ingestion at baseline and after 4 weeks of supplementation.
Change in microvascular endothelial function in the fasted condition | 4 weeks
  Microvascular endothelial function will be assessed using peripheral arterial tonometry (EndoPAT device) during reactive hyperemia at baseline and after 4 weeks of supplementation.
Change in microvascular endothelial function in the fasted condition | 4 weeks
  Microvascular endothelial function will be assessed using forearm muscle oxygenation (near-infrared spectroscopy) during reactive hyperemia at baseline and after 4 weeks of supplementation.
Change in microvascular endothelial function during acute hyperglycemia | 4 weeks
  Microvascular endothelial function will be assessed using forearm muscle oxygenation (near-infrared spectroscopy) during reactive hyperemia at 60 minutes after oral glucose ingestion at baseline and after 4 weeks of supplementation.
Change in blood glucose levels in the fasted condition | 4 weeks
  Blood glucose levels will be measured by finger prick at baseline and after 4 weeks of supplementation.
Change in blood glucose levels during acute hyperglycemia | 4 weeks
  Blood glucose levels will be measured by finger prick at 60 minutes after oral glucose ingestion at baseline and after 4 weeks of supplementation.
Change in central and peripheral arterial stiffness in the fasted condition | 4 weeks
  Arterial stiffness will be assessed using the central (carotid-femoral) and peripheral (femoral-ankle) pulse wave velocity at baseline and after 4 weeks of supplementation.
Change in central and peripheral arterial stiffness during acute hyperglycemia | 4 weeks
  Arterial stiffness will be assessed using the central (carotid-femoral) and peripheral (femoral-ankle) pulse wave velocity at 60 minutes after oral glucose ingestion at baseline and after 4 weeks of supplementation.
Change in blood pressure in the fasted condition | 4 weeks
  Brachial and aortic blood pressure will be measured using an automated sphygmomanometry arm cuff (SphygmoCor XCEL). Beat-to-beat blood pressure will be measured using an automated photoplethysmography finger cuff (Finometer). Blood pressure will be measured at baseline and after 4 weeks of supplementation.
Change in blood pressure during acute hyperglycemia | 4 weeks
  Brachial and aortic blood pressure will be measured using an automated sphygmomanometry arm cuff (SphygmoCor XCEL). Beat-to-beat blood pressure will be measured using an automated photoplethysmography finger cuff (Finometer). Blood pressure will be measured at 60 minutes after oral glucose ingestion at baseline and after 4 weeks of supplementation.
Change in stroke volume in the fasted condition | 4 weeks
  Stroke volume will be measured using impedance cardiography (PhysioFlow) at baseline and after 4 weeks of supplementation.
Change in stroke volume during acute hyperglycemia | 4 weeks
  Stroke volume will be measured using impedance cardiography (PhysioFlow) at 60 minutes after oral glucose ingestion at baseline and after 4 weeks of supplementation.
Change in total peripheral resistance in the fasted condition | 4 weeks
  Total peripheral resistance will be measured using impedance cardiography (PhysioFlow) at baseline and after 4 weeks of supplementation.
Change in total peripheral resistance during acute hyperglycemia | 4 weeks
  Total peripheral resistance will be measured using impedance cardiography (PhysioFlow) at 60 minutes after oral glucose ingestion at baseline and after 4 weeks of supplementation.

SECONDARY OUTCOMES:
Change in body composition | 4 weeks
  Body composition (fat and lean mass) will be measured at baseline and after 4 weeks of supplementation.
Change in muscle strength | 4 weeks
  Maximal handgrip strength will be measured using handgrip dynamometer. Leg extension and plantar flexion strength will be measured using the 10RM test at baseline and after 4 weeks of supplementation.
Change in insulin levels | 4 weeks
  Serum insulin levels will be tested at baseline and after 4 weeks of supplementation.
Change in serum arginine levels | 4 weeks
  Serum arginine levels will tested at baseline and after 4 weeks of supplementation.
Change in serum arginase activity levels | 4 weeks
  Serum arginase activity levels will tested at baseline and after 4 weeks of supplementation.
Change in 24-hour ambulatory blood pressure monitoring | 4 weeks
  Ambulatory blood pressure will be obtained using a monitor during daytime and nighttime on two separate days at baseline and after 4 weeks of supplementation.

CONTACTS AND LOCATIONS:
Overall Officials: Arturo Figueroa, Ph.D, MD, Principal Investigator — Texas Tech University
Locations (1):
- TTU Kinesiology and Sport Management Building, Lubbock, Texas, United States

IPD SHARING:
Plan to Share IPD: No